CLINICAL TRIAL: NCT01109277
Title: An Evidence-based Strategy for Assessing the Risk of Significant Neonatal Hyperbilirubinemia
Brief Title: Prediction of Neonatal Hyperbilirubinemia
Acronym: 2010ICTPAGR
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Fouzas Sotirios, Neonatal Intensive Care Unit, Department of Pediatrics, University Hospital of Patras
Other Study IDs: 2010ICTPAGR
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2010-04

CONDITIONS: Hyperbilirubinemia, Neonatal
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy term and late-preterm neonates

SUMMARY:
Objective: To develop an evidence-based strategy for assessing the risk of significant hyperbilirubinemia in healthy term and near-term (late-preterm) neonates.

Hypothesis: A stepwise strategy which combines clinical parameters and serial non-invasive transcutaneous bilirubin (TcB) values could reliably predict significant neonatal hyperbilirubinemia.

Methods: Data from neonates >34 weeks' gestation included in the registry for neonatal hyperbilirubinemia of the well-baby nursery of the University Hospital of Patras, from January 2008 to December 2010 will be reviewed.

The registry includes prospectively collected data such as sex, gestational age, gestation and perinatal information, mother's and infant's ABO group and Rh, G6PD deficiency, Coombs test, type of delivery and complications, birthweight, postnatal medications and interventions, type and volume of feeding (daily), extension of jaundice, TcB measurements at intervals of 12+/-4 hours until discharge, total serum bilirubin values (if obtained), TcB or TSB measurements at follow-up, weight at discharge, need of phototherapy (inpatient or after discharge). TcB and TSB values are plotted on a hour-specific chart.

A novel predictive nomogram based on TcB measurements (Varvarigou et al. Pediatrics 2009;124:1052-9) will be used to classify TcB values as high, intermediate, and low risk.

Significant hyperbilirubinemia will be defined as a TSB value above the phototherapy threshold level according to the AAP 2004 guidelines

Statistics: Independent and joint effects of various clinical factors on the development of significant hyperbilirubinemia will be evaluated by logistic regression analysis Cluster analysis and Chi-squared Automatic Interaction Detection (CHAID) tree method will be used to develop the strategy. At each step, CHAID chooses the independent (predictor) variable that has the strongest interaction with the dependent variable. Categories of each predictor are merged if they are not significantly different with respect to the dependent variable.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term and late-preterm neonates

Exclusion Criteria:

* Admission to the NICU

Ages: 1 Hour to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy term and late-preterm neonates
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Risk of significant hyperbilirubinemia assessed by an evidence-based strategy | Birth to 14th postnatal day
  Risk for significant hyperbilirubinemia (defined as serum bilirubin values above the phototherapy threshold according to the American Academy of Pediatrics 2004 guidelines) assessed by a strategy which will combine clinical risk factors and non-invasive TcB measurements

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Varvarigou, Prof, Study Director — Neonatal Intensive Care Unit, Department of Pediatrics, University Hospital of Patras; Sotirios Fouzas, MD, Principal Investigator — Neonatal Intensive Care Unit, University Hospital of Patras; Aggeliki Karatza, MD, Principal Investigator — Neonatal Intensive Care Unit, University Hospital of Patras; Lito Mantagou, MD, Principal Investigator — Pediatric Department, University Hospital of Patras
Locations (1):
- Well-baby nursery, Department of Pediatrics, University Hospital of Patras, Pátrai, Greece